CLINICAL TRIAL: NCT04632251
Title: Evaluation of the SENSEI® Laparoscopic Tethered Gamma Probe for 99mTc-nanocolloid Sentinel Lymph Node Biopsy in Prostate Cancer
Acronym: LPM-012
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lightpoint Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LPM-012
Record Dates: First submitted 2020-09-21; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Familiarisation (Other): The first 2 patients per site (N = 10 in total) are considered to be sufficient to enable further familiarisation with the procedure and use of the probe in addition to the usability work and training that the sites did prior to the start of this study.
  Interventions: Device: SENSEI®

INTERVENTIONS:
Device: SENSEI® — SENSEI® laparoscopic tethered gamma probe is an intra-operative laparoscopic gamma probe system

SUMMARY:
This study is a prospective, open label, single-arm study to examine the performance and safety of the SENSEI® laparoscopic tethered gamma probe in patients undergoing 99mTc-nanocolloid SLNB for prostate cancer (PCa) during RP and ePLND surgery.

Patients scheduled for RP and ePLND using the standard treatment pathways at each centre will have preoperative 99mTc-nanocolloid imaging. RP and ePLND will be conducted as standard of care, with SLNB guided by the SENSEI® laparoscopic tethered gamma probe carried out after RP and prior to ePLND. The first 2 patients per site (N = 10 in total) are considered to be sufficient to enable further familiarisation with the procedure and use of the probe in addition to the usability work and training that the sites did prior to the start of this study. Subsequent patients will be evaluable for the PP population. The primary analysis of diagnostic performance will be performed using the PP population of patients with SLN identified on preoperative imaging

ELIGIBILITY:
Inclusion Criteria:

* Male subjects who are ≥ 18 years of age with histologically proven prostate cancer; and who have signed an informed consent form prior to any study related activity • Subjects who are scheduled for radical prostatectomy with ePLND.

Exclusion Criteria:

* Subjects who have received prior prostate cancer treatment or prior pelvic surgery;

  * Subjects who have an existing medical condition that would compromise their participation in the study;
  * Subjects with a history of hypersensitivity to 99mTc-nanocolloid or any excipients;
  * Subjects who are unable to give voluntary, written informed consent to participate in this study;
  * Subjects who are unable to understand this study and are not willing to complete all the study assessments.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 56 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-02-16 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Sentinel lymph node (SLN) detection rate with the SENSEI® laparoscopic tethered gamma probe. Detection rate is defined as the percentage of patients with at least one SLN detected intraoperatively. | Length of study finish - 6 Months

SECONDARY OUTCOMES:
Number of SLNs detected with the SENSEI® laparoscopic tethered gamma probe in comparison to preoperative planar LS and SPECT/CT in centres with a SPECT/CT scanner. | Length of study finish - 6 Months
Diagnostic performance of the SENSEI® laparoscopic tethered gamma probe for detecting SLNs | Length of study finish - 6 Months
  Diagnostic performance include sensitivity, specificity, accuracy, positive predictive value (PPV) and negative predictive value (NPV). Histopathological tumour status of lymph nodes excised based on the ePLND template will be used as reference standard.
Overall ease of use of the SENSEI® laparoscopic tethered gamma probe. | Length of study finish - 6 Months
Radiation safety measurements for the staff. | Length of study finish - 6 Months
Duration of surgery | Length of study finish - 6 Months
  Outcome will be measured from the first skin incision to skin closure (skin to skin).
In centres using a conventional rigid laparoscopic gamma probe: | Length of study finish - 6 Months
  SLN detection rate, number of SLNs, diagnostic performance and in vivo and ex vivo count rate of the SENSEI® laparoscopic tethered gamma probe in comparison to the conventional rigid laparoscopic gamma probe.
  In centres using a conventional rigid laparoscopic gamma probe: Overall ease of use of the conventional rigid laparoscopic gamma probe
Comparison of detection rates between robotic, open and manual laparoscopic surgery | Length of study finish - 6 Months
Incidence of study-related Adverse Events | Length of study finish - 6 Months
Complication rate as measured by Clavien-Dindo classification | Length of study finish - 6 Months
In centres using a conventional rigid laparoscopic gamma probe: Overall ease of use of the conventional rigid laparoscopic gamma probe | Length of study finish - 6 Months
  Outcome will be assessed using questionnaire and ethnographic observations, and at similar time points.
Duration of Sentinel Lymph Node Biopsy separately for each probe used | Length of study finish - 6 Months
  Duration of SLNB will be measured from the first in vivo measurement to completion of ex vivo measurements of excised SLN specimens and measured separately for each probe used. The end time of ex vivo measurements of the excised ePLND specimens will also be recorded.
Sentinel Lymph Node detection Rate | Length of study finish - 6 Months
  The 95% Confidence Interval (CI) around the detection rate will allow an estimate of the true detection rate. The sample size directly impacts the precision of the estimate. The sample size of 40 evaluable patients has been selected to provide a reasonable level of precision for the estimate of the SLN detection rate
Number of Sentinel Lymph Nodes | Length of study finish - 6 Months
  Number of SLNs detected with the SENSEI® laparoscopic tethered gamma probe in comparison to preoperative planar LS and SPECT/CT in centres with a SPECT/CT scanner.
Diagnostic performance and in vivo and ex vivo count rate of the SENSEI® laparoscopic tethered gamma probe in comparison to the conventional rigid laparoscopic gamma probe. | Length of study finish - 6 Months

CONTACTS AND LOCATIONS:
Locations (4):
- UZ Leuven, Leuven, Belgium
- Institute Paoli-Calmettes, Marseille, France
- University Hospital Essen, Essen, Germany
- Hospital del Mar, Barcelona, Spain

REFERENCES:
- [Derived] Abascal Junquera JM, Harke NN, Walz JC, Hadaschik B, Adshead J, Everaerts W, Goffin K, Grootendorst MR, Oldfield F, Vyas K, Fusco AM, Juanpere N, Vidal-Sicart S, Fumado L. A Drop-in Gamma Probe for Minimally Invasive Sentinel Lymph Node Dissection in Prostate Cancer: Preclinical Evaluation and Interim Results From a Multicenter Clinical Trial. Clin Nucl Med. 2023 Mar 1;48(3):213-220. doi: 10.1097/RLU.0000000000004557. Epub 2023 Jan 14. PMID 36723880